CLINICAL TRIAL: NCT00481702
Title: A Prospective, Multicenter, Open-Label, Randomized, Comparative Study to Evaluate the Efficacy, Safety, and Tolerability of Ertapenem Versus Ceftriaxone/Metronidazole in the Treatment of Intra-Abdominal Infections in Adults
Brief Title: A Study to Evaluate the Safety and Effectiveness of Ertapenem Versus Ceftriaxone/Metronidazole in the Treatment of Intra-abdominal Infections in Adults (0826-802)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0826-802; 2007_558
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Intra-abdominal Infection
MeSH Terms: conditions — Intraabdominal Infections | interventions — Duration of Therapy; Ertapenem

INTERVENTIONS:
Drug: Comparator: ceftriaxone sodium / Duration of Treatment: 8 Weeks
Drug: MK0826, /Duration of Treatment : 8 Weeks
Drug: Comparator: metronidazole / Duration of Treatment: 8 Weeks

SUMMARY:
A multicenter study to evaluate the effectiveness of ertapenem compared to ceftriaxone/metronidazole in treating certain abdominal infections that require surgery in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age 18 or older
* Patient has a diagnosis of intra-abdominal infection requiring surgery as evidenced by fever, elevated while blood cell count and abdominal pain

Exclusion Criteria:

* Patient has another infection, other than abdominal
* Female patient is pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-12; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
That ertapenem is as effective as ceftriaxone/metronidazole in the treatment of an abdominal infection | 2 weeks after treatment

SECONDARY OUTCOMES:
That ertapenem is as effective as ceftriaxone/metronidazole in the treatment of abdominal infection | 4 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Navarro NS Jr, Campos MI, Alvarado R, Quintero N, Branicki FJ, Wei J, Shivaprakash M, Vrijens F, Giezek H, Chan CY, DiNubile MJ; Oasis II Study Team. Ertapenem versus ceftriaxone and metronidazole as treatment for complicated intra-abdominal infections. Int J Surg. 2005;3(1):25-34. doi: 10.1016/j.ijsu.2005.03.010. PMID 17462256
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html